CLINICAL TRIAL: NCT01349868
Title: A Randomized, Double-Blind, Single Dose, Six-Treatment, Placebo-Controlled, Cross-Over, Multi-Center Study to Assess Efficacy and Safety of Three Doses of PT005, in Patients With Moderate to Severe COPD, Compared With Foradil® Aerolizer® (12 and 24 µg Open-Label) as Active Controls
Brief Title: PT005 MDI Dose Ranging Versus Foradil Aerolizer Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT005003
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PT005 MDI (Dose 1) (Experimental): PT005 MDI (Dose 1)
  Interventions: Drug: PT005 MDI
- PT005 MDI (Dose 2) (Experimental): PT005 MDI (Dose 2)
  Interventions: Drug: PT005 MDI
- PT005 MDI (Dose 3) (Experimental): PT005 MDI (Dose 3)
  Interventions: Drug: PT005 MDI
- Placebo MDI (Placebo Comparator): Placebo MDI
  Interventions: Other: Placebo MDI
- Formoterol Fumarate 12 μg (Foradil® Aerolizer®) (Active Comparator): Formoterol fumarate inhalation powder 12 μg
  Interventions: Drug: Formoterol Fumarate 12 μg (Foradil® Aerolizer®)
- Formoterol Fumarate 24 μg (Foradil® Aerolizer®) (Active Comparator): Formoterol fumarate inhalation powder 24 μg
  Interventions: Drug: Formoterol Fumarate 24 μg (Foradil® Aerolizer®)

INTERVENTIONS:
Drug: PT005 MDI — PT005 MDI taken as two inhalations
  Arms: PT005 MDI (Dose 1); PT005 MDI (Dose 2); PT005 MDI (Dose 3)
Drug: Formoterol Fumarate 12 μg (Foradil® Aerolizer®) — Taken as 1 capsule. Each capsule contains 12 μg corresponding to 10 µg formoterol fumarate dihydrate delivered from the mouthpiece
  Other Names: Foradil® Aerolizer®
  Arms: Formoterol Fumarate 12 μg (Foradil® Aerolizer®)
Drug: Formoterol Fumarate 24 μg (Foradil® Aerolizer®) — Taken as 2 capsules. Each capsule contains 12 μg corresponding to 10 µg formoterol fumarate dihydrate delivered from the mouthpiece
  Other Names: Foradil® Aerolizer®
  Arms: Formoterol Fumarate 24 μg (Foradil® Aerolizer®)
Other: Placebo MDI — Matching placebo to PT005 MDI taken as two inhalations
  Arms: Placebo MDI

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of inhaled PT005 MDI compared to placebo and Foradil Aerolizer in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Clinical history of COPD with airflow limitation that is not fully reversible
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post- bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post- bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Able to change COPD treatment as required by protocol
* Demonstratead reversibility to short acting beta agonist (Ventolin HFA) (> 12% and >150 mL improvement in baseline FEV1 approximately 30 minutes following administration of 4 puffs of Ventolin HFA or > 200 mL improvement in baseline FEV1 30 minutes following administration of 2 puffs of Ventolin HFA)

Key Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 3 months of Screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG, uncontrolled hypertension, glaucoma, symptomatic prostatic hypertrophy)
* Cancer that has not been in complete remission for at least 5 years
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives

Other inclusion/exclusion criteria as defined by the protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 AUC0-12 from test day baseline across the three doses of inhaled PT005 compared with placebo | 1 Day
  The primary objective of this study is to demonstrate efficacy relative to placebo of PT005 MDI in patients with moderate to severe chronic obstructive pulmonary disease (COPD) within the range of doses evaluated in this study. To this end, each dose of PT005 MDI will be compared to placebo with respect to the primary efficacy endpoint, the change in FEV1 AUC0-12 from baseline.

SECONDARY OUTCOMES:
Characterize the dose-response curve of PT005 MDI | 1 Day
  The secondary objective of the study is to characterize the dose-response curve of PT005 MDI, to conduct a non-inferiority assessment comparing PT005 MDI within the range of doses evaluated in this study to open-label Foradil Aerolizer 12 µg, and to select the most appropriate dose of PT005 MDI to carry forward into Phase III clinical studies
Safety measures including electrocardiograms (ECGs), vital signs, physical exam, clinical laboratory testing, and adverse events | 1 Day

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Tampa, Florida
  - Pearl Investigative Site, Spartanburg, South Carolina